CLINICAL TRIAL: NCT01154478
Title: Effects of Polyphenols and Omega-3 Fatty Acids on Cardiovascular Rik Factors (Focusing on Postprandial Lipids Metabolism) in Subjects With High Risk for Type 2 Diabetes and Cardiovascular Diseases
Brief Title: Effects of Dietary Polyphenols and ω-3 Fatty Acids on Cardiovascular Risk Factors in High Risk Subjects
Acronym: Etherpaths
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Associate Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EpWP5
Record Dates: First submitted 2010-06-14; First posted 2010-07-01 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Metabolic Syndrome
Keywords: polyphenols omega-3 postprandial lipemia adipose tissue
MeSH Terms: conditions — Metabolic Syndrome | interventions — Fatty Acids, Omega-3; Polyphenols; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- B group (Experimental): Diet rich in omega-3 fatty acids
  Interventions: Other: Diet rich in omega-3 fatty acids
- C group (Experimental): Diet rich in polyphenols
  Interventions: Other: Diet rich in polyphenols
- D group (Experimental): Diet rich in polyphenols and in omega-3 fatty acids
  Interventions: Other: diet rich in omega-3 and polyphenols
- A group (control group) (Placebo Comparator): diet with low content of omega-3 fatty acids and polyphenols
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Diet rich in omega-3 fatty acids — fish at least 3 times per week, large leaf vegetables
  Arms: B group
Other: Diet rich in polyphenols — extra virgin olive oil, green tea, berries,fruits rich in polyphenols, dark chocolate, decaffenated coffee
  Arms: C group
Other: Control diet — low content of omega-3 fatty acids and polyphenols (low intake of fish, nuts and legumes,oil rich in monounsaturated fatty acids, vegetables and fruits poor in polyphenols)
  Arms: A group (control group)
Other: diet rich in omega-3 and polyphenols — Fish at least 3 times x week,large leaf vegetables + extra virgin olive oil, green tea, berries,fruits rich in polyphenols, dark chocolate, decaffenated coffee
  Arms: D group

SUMMARY:
The aim of this study is to explore if a 8-weeks dietary intervention with polyphenols and omega 3 fatty acids (alone or combined) may be effective on postprandial lipids metabolism and other cardiovascular risk factors in people at high cardiovascular risk.

DETAILED DESCRIPTION:
Fish consumption is associated with a lower cardiovascular risk and dietary supplementation with ω-3 fatty acids reduces plasma triglyceride levels. The mechanisms of action of ω-3 fatty acids are currently not completely understood. It has been hypothesized that polyunsaturated ω-3 fatty acids beneficial effects may be mediated through their ability to facilitate plasmalogen replenishment.

Polyphenols are associated with beneficial effects on some cardiovascular risk factors, in particular with a reduced lipid oxidation. Less data are available on their effects on lipid metabolism. Recent data suggest that these effects could be mediated by changes in plasmalogen levels.

The effects on lipid metabolism of combining the two dietary approaches (ω-3 fatty acids and polyphenols) are not known.

While developed populations live for the most part in the postprandial state, much of the information on lipid metabolism refers to fasting condition.

Dietary Intervention Study Design

Eighty people at high cardiovascular risk randomly assigned to one of the four different nutritional 8-week interventions:

(A) Control diet poor in omega-3 fatty acids and polyphenols (B) Diet rich in omega-3 fatty acids (C) Diet rich in polyphenols (D) Diet rich in omega-3 fatty acids and polyphenols

ELIGIBILITY:
Inclusion Criteria:

* bmi >25<35 kg/m2
* High waist circumference (men >102 cm, women >88 cm) + one the following components of metabolic syndrome :

Fasting plasma triglycerides ≥150 mg/dl Fasting HDL-col <40 mg/dl (men) and <50 mg/dl (women) Fasting plasma glucose 100-125 mg/dl

Exclusion Criteria:

* Fasting plasma triglycerides ≥400 mg/dl and cholesterol >270 mg/dl
* Cardiovascular events (AMI and/or stroke) in the last 6 months
* Diabetes mellitus
* Regular intensive physical activity
* Kidney (serum creatinine >1.7 mg/dl) and liver (transaminases >double)
* Hypolipidemic or antinflammatory drugs
* Anemia (Hb <12 g/dl) or any other chronic disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
incremental AUC after a test meal of triglycerides concentration in chylomicrons and VLDL fraction | 48 months

SECONDARY OUTCOMES:
insulin sensitivity | 48 months
plasma and adipose tissue adipokines | 48 months
endothelial function | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Annuzzi, Study Director — Federico II University
Locations (1):
- Federico II University, Napoli, Naples, Italy

REFERENCES:
- [Derived] Costabile G, Vetrani C, Bozzetto L, Giacco R, Bresciani L, Del Rio D, Vitale M, Della Pepa G, Brighenti F, Riccardi G, Rivellese AA, Annuzzi G. Plasma TMAO increase after healthy diets: results from 2 randomized controlled trials with dietary fish, polyphenols, and whole-grain cereals. Am J Clin Nutr. 2021 Oct 4;114(4):1342-1350. doi: 10.1093/ajcn/nqab188. PMID 34091663
- [Derived] Della Pepa G, Vetrani C, Vitale M, Bozzetto L, Costabile G, Cipriano P, Mangione A, Patti L, Riccardi G, Rivellese AA, Annuzzi G. Effects of a diet naturally rich in polyphenols on lipid composition of postprandial lipoproteins in high cardiometabolic risk individuals: an ancillary analysis of a randomized controlled trial. Eur J Clin Nutr. 2020 Jan;74(1):183-192. doi: 10.1038/s41430-019-0459-0. Epub 2019 Jun 27. PMID 31249395
- [Derived] Bozzetto L, Annuzzi G, Ragucci M, Di Donato O, Della Pepa G, Della Corte G, Griffo E, Anniballi G, Giacco A, Mancini M, Rivellese AA. Insulin resistance, postprandial GLP-1 and adaptive immunity are the main predictors of NAFLD in a homogeneous population at high cardiovascular risk. Nutr Metab Cardiovasc Dis. 2016 Jul;26(7):623-629. doi: 10.1016/j.numecd.2016.01.011. Epub 2016 Apr 14. PMID 27134062
- [Derived] Bozzetto L, Annuzzi G, Pacini G, Costabile G, Vetrani C, Vitale M, Griffo E, Giacco A, De Natale C, Cocozza S, Della Pepa G, Tura A, Riccardi G, Rivellese AA. Polyphenol-rich diets improve glucose metabolism in people at high cardiometabolic risk: a controlled randomised intervention trial. Diabetologia. 2015 Jul;58(7):1551-60. doi: 10.1007/s00125-015-3592-x. Epub 2015 Apr 24. PMID 25906754